CLINICAL TRIAL: NCT03040141
Title: Phase 2b, Multicenter, Randomized, Double-blind Study to Evaluate the Efficacy and Safety of IV VIS410 in Addition to Oseltamivir Compared With Oseltamivir Alone in Hospitalized Adults With Influenza A Infection Requiring Oxygen Support
Brief Title: Study of Efficacy and Safety of IV VIS410 Plus Oseltamivir Versus Oseltamivir in Hospitalized Adults With Influenza A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Visterra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIS410-203
Record Dates: First submitted 2017-01-23; First posted 2017-02-02 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Influenza A
MeSH Terms: interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VIS410 low dose (Experimental): Single intravenous infusion of fixed low dose of VIS410 in addition to oseltamivir
  Interventions: Drug: Low dose of VIS410
- VIS410 high dose (Experimental): Single intravenous infusion of fixed high dose of VIS410 in addition to oseltamivir
  Interventions: Drug: High dose of VIS410
- Placebo (Placebo Comparator): Single intravenous infusion of placebo in addition to oseltamivir
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose of VIS410 — Single intravenous infusion of fixed low dose of VIS410 in addition to oseltamivir
  Other Names: oseltamivir
  Arms: VIS410 low dose
Drug: High dose of VIS410 — Single intravenous infusion of fixed high dose of VIS410 in addition to oseltamivir
  Other Names: oseltamivir
  Arms: VIS410 high dose
Drug: Placebo — Single intravenous infusion of placebo in addition to oseltamivir
  Other Names: oseltamivir
  Arms: Placebo

SUMMARY:
This study is to compare the efficacy and safety of VIS410 in combination with oseltamivir vs oseltamivir alone in severely ill subjects with influenza A infection requiring oxygen support.

DETAILED DESCRIPTION:
This study is to compare the efficacy and safety of VIS410 in combination with oseltamivir vs oseltamivir alone in severely ill subjects with influenza A infection requiring oxygen support. Subjects will be followed for 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥ 18 years.
* Test positive for influenza A by rapid antigen test or with another commercially available test on an adequate nasopharyngeal specimen in accordance with the manufacturer's instructions, or an acceptable local test, including PCR (Polymerase chain reaction), FIA (Fluorescent immunoassay), or ELISA
* Onset of influenza symptoms no more than 5 days before VIS410/placebo infusion; symptoms may include cough, dyspnea, sore throat, fever, myalgias, headache, nasal symptoms (rhinorrhea, congestion), fatigue, diarrhea, anorexia, nausea, and vomiting.
* Requirement for oxygen support including any positive pressure ventilation
* Women of childbearing potential must have a negative pregnancy test within 2 days prior to VIS410/placebo infusion.
* Women should fulfill one of the following criteria:

  * Post-menopausal; either amenorrhea ≥ 12 months or follicle stimulating hormone > 40 mIU/mL as documented in their medical history
  * Surgically sterile; hysterectomy, bilateral oophorectomy, or tubal ligation
  * Women of childbearing potential participating in heterosexual sexual relations must be willing to use adequate contraception from screening until 60 days post VIS410/placebo infusion.
* Non-vasectomized (or vasectomized less than 6 months prior to dosing) male subjects who have a female partner of childbearing potential must use an effective birth control method from screening until 60 days post VIS410/placebo infusion.
* Subject, or a legally acceptable representative (LAR), is able to understand the purpose and risks of the study and willing to give voluntary written informed consent.

Exclusion Criteria:

* Known or suspected intolerance or hypersensitivity to VIS410, oseltamivir, pretreatment medications (diphenhydramine, or to both ibuprofen and acetylsalicylic acid [ASA]), or closely related compounds (eg, other monoclonal antibodies)
* Subjects who have received VIS410 in the past
* History of receiving monoclonal antibody products (including VIS410) within 3 months prior to VIS410/placebo dosing or planned administration during the study period
* Subjects who have taken more than 6 doses of an approved antiviral therapy for influenza within the prior 96 hours (eg, oral oseltamivir, inhaled zanamivir, IV peramivir, or oral ribavirin) between onset of symptoms and VIS410/placebo dosing
* Subjects with known co-infection with influenza B or other viral respiratory infections (e.g., respiratory syncytial virus, parainfluenza viruses, respiratory adenoviruses)
* Subjects with lung transplant or history of severe chronic lung disease, including cystic fibrosis or any condition requiring home oxygen therapy
* Subjects on extracorporeal membrane oxygenation (ECMO) at time of randomization
* Subjects with end stage renal disease who are not undergoing hemodialysis
* Subjects with active graft-vs-host disease, hematopoietic stem cell transplant within the previous 90 days, or human immunodeficiency virus infection with a CD4 cell count of less than 200 per cubic millimeter
* Hospitalization for > 48 hours prior to randomization
* High probability of mortality within 48 hours of randomization as determined by the Investigator
* Subjects weighing less than 45 kg
* Enrollment in any other investigational drug or device study, any disease or vaccine study within 30 days prior to Day 1 or within 5 half-lives of the investigational compound, whichever is longer
* Known or suspected alcohol or drug abuse, that is, abuse of a level that would compromise the safety or cooperation of the subject in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Oldach, MD, Principal Investigator — Visterra, Inc.
Locations (101):
- United States (21):
  - Visterra, Tucson, Arizona
  - Visterra, Stanford, California
  - Visterra, St. Petersburg, Florida
  - Visterra, Atlanta, Georgia
  - Visterra, Decatur, Georgia
  - Visterra, Blackfoot, Idaho
  - Visterra, Chicago, Illinois
  - Visterra, Detroit, Michigan
  - Visterra, Butte, Montana
  - Visterra, Albany, New York
  - Visterra, Syracuse, New York
  - Visterra, Durham, North Carolina
  - Visterra, Greensboro, North Carolina
  - Visterra, Cleveland, Ohio
  - Visterra, Columbus, Ohio
  - Visterra, Allentown, Pennsylvania
  - Visterra, Philadelphia, Pennsylvania
  - Visterra, York, Pennsylvania
  - Visterra, Roanoke, Virginia
  - Visterra, Richland, Washington
  - Visterra, Tacoma, Washington
- Australia (6):
  - Visterra, Adelaide, South Australia
  - Visterra, Melbourne
  - Visterra, Parkville
  - Visterra, South Brisbane
  - Visterra, Westmead
  - Visterra, Woolloongabba
- Belarus (6):
  - Visterra, Brest
  - Visterra, Grodno
  - Visterra, Homyel
  - Visterra, Lesnoy
  - Visterra, Minsk
  - Visterra, Vitebsk
- Belgium (2):
  - Visterra, Brussels
  - Visterra, Edegem
- Bulgaria (5):
  - Visterra, Kozloduy
  - Visterra, Montana
  - Visterra, Plovdiv
  - Visterra, Sofia
  - Visterra, Veliko Tarnovo
- Visterra, Moncton, New Brunswick, Canada
- Estonia (3):
  - Visterra, Pärnu
  - Visterra, Tallinn
  - Visterra, Tartu
- France (7):
  - Visterra, La Roche-sur-Yon
  - Visterra, La Tronche
  - Visterra, Limoges
  - Visterra, Metz-Tessy
  - Visterra, Nantes
  - Visterra, Paris
  - Visterra, Quimper
- Visterra, Tbilisi, Georgia
- Latvia (6):
  - Visterra, Daugavpils
  - Visterra, Liepāja
  - Visterra, Rēzekne
  - Visterra, Riga
  - Visterra, Valmiera
  - Visterra, Ventspils
- Malaysia (3):
  - Visterra, Alor Star, Kedah
  - Visterra, Kuala Lumpur, Kuala Lumpur
  - Visterra, Taiping, Perak
- New Zealand (2):
  - Visterra, Auckland
  - Visterra, Wellington
- Russia (6):
  - Visterra, Arkhangelsk
  - Visterra, Kazan'
  - Visterra, Novosibirsk
  - Visterra, Smolensk
  - Visterra, Tomsk
  - Visterra, Vladimir
- Serbia (3):
  - Visterra, Kragujevac
  - Visterra, Niš
  - Visterra, Novi Sad
- Visterra, Singapore, Singapore
- South Africa (8):
  - Visterra, Lyttelton, Centurion
  - Visterra, Auckland Park, Gauteng
  - Visterra, Pretoria, Gauteng
  - Visterra, Thabazimbi, Limpopo
  - Visterra, Benoni
  - Visterra, Cape Town
  - Visterra, Durban
  - Visterra, Worcester
- Spain (8):
  - Visterra, Alicante
  - Visterra, Badalona
  - Visterra, Barakaldo
  - Visterra, Barcelona
  - Visterra, Córdoba
  - Visterra, Granada
  - Visterra, Madrid
  - Visterra, Terrassa
- Thailand (3):
  - Visterra, Bangkok
  - Visterra, Khon Kaen
  - Visterra, Nonthaburi
- Turkey (Türkiye) (3):
  - Visterra, Ankara
  - Visterra, Istanbul
  - Visterra, Trabzon
- Ukraine (6):
  - Visterra, Ivano-Frankivsk
  - Visterra, Kyiv
  - Visterra, Odesa
  - Visterra, Poltava
  - Visterra, Sumy
  - Visterra, Zhytomyr

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Approximately 120 participants were planned however, a total of 89 subjects were randomized to treatment. 73 participants completed the trial. There were study discontinuations for death, consent withdrawn and participants who were enrolled, but did not receive study drug.
Groups:
- VIS410 High Dose: VIS410 liquid for infusion. Single, fixed, intravenous dose of 4000 mg in addition to oseltamivir
- VIS410 Low Dose: VIS410 liquid for infusion. Single, fixed, intravenous dose of 2000 mg in addition to oseltamivir
Period: Overall Study
Arm/Group | VIS410 High Dose | VIS410 Low Dose | Placebo
Started | 29 | 30 | 30
Completed | 25 | 24 | 24
Not Completed | 4 | 6 | 6
Not completed — Death | 1 | 2 | 3
Not completed — Withdrawal by Subject | 3 | 1 | 1
Not completed — Subject discharged to nursing home, not able to attend visits | 0 | 1 | 0
Not completed — Subject did not receive study drug or was not confirmed Influenza A positive | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Modified Intent to treat (MITT) population. All subjects of the safety population that have an assessment of O2 support after randomization and are confirmed influenza A positive. Subjects will be analyzed based on the treatment to which they were randomized, irrespective of what they actually received. This population was selected for the analysis of the primary endpoint to maintain the benefits of randomization and avoid the bias associated with the non-random loss of the participants
Groups:
- Total: Total of all reporting groups
Arm/Group | VIS410 High Dose | VIS410 Low Dose | Placebo | Total
Number analyzed (Participants) | 29 | 28 | 28 | 85
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age (years) | 60 (19.00) | 66.2 (13.94) | 57.5 (22.41) | 61.2 (18.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 13 | 44
  Male | 16 | 10 | 15 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 00 | 3 | 5
  Not Hispanic or Latino | 27 | 28 | 24 | 79
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 1 | 4
  White | 25 | 17 | 19 | 61
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 5 | 14
Region of Enrollment [Number; unit: participants]
  Singapore | 0 | 0 | 1 | 1
  United States | 3 | 4 | 2 | 9
  Malaysia | 1 | 0 | 1 | 2
  Belarus | 1 | 0 | 0 | 1
  Thailand | 3 | 6 | 2 | 11
  Spain | 4 | 4 | 4 | 12
  Latvia | 2 | 1 | 3 | 6
  Belgium | 0 | 0 | 2 | 2
  South Africa | 2 | 1 | 3 | 6
  Georgia | 0 | 1 | 0 | 1
  Bulgaria | 3 | 0 | 1 | 4
  France | 1 | 2 | 2 | 5
  Serbia | 6 | 5 | 3 | 14
  Australia | 0 | 1 | 1 | 2
  Estonia | 3 | 3 | 3 | 9
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: Kg/m^2] | 28.2 (6.48) | 28.4 (7.93) | 29.2 (6.3) | 28.6 (6.87)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Status of Participants on Day 7
Description: Evaluate the effect of 2 dose levels of VIS410 + oseltamivir on clinical status using a seven-level ordinal scale. Comparison between treatment groups and between all VIS410 recipients versus placebo were assessed.
Time Frame: 7 days
Population: Modified Intent to treat (MITT) population. All participants of the safety population that have an assessment of O2 support after randomization and are confirmed influenza A positive. Participants will be analyzed based on the treatment to which they were randomized, irrespective of what they actually received. This population was selected for the analysis of the primary endpoint to maintain the benefits of randomization and avoid the bias associated with the non-random loss of the participants
Measure: Count of Participants; unit: Participants
Groups:
- VIS410 Total: Combined results from VIS410 high and low dose groups
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 28 | 57 | 28
Participants
  Death | 1 | 1 | 2 | 1
  ICU stay with mechanical ventilation | 1 | 2 | 3 | 1
  ICU stay without mechanical ventilation | 2 | 0 | 2 | 0
  Non-ICU hospitalization with supplemental oxygen | 5 | 5 | 10 | 3
  Non-ICU hospitalization without supplemental oxygen | 12 | 8 | 20 | 10
  Discharge with partial resumption of normal activities | 7 | 5 | 12 | 11
  Discharge with full resumption of normal activities | 1 | 7 | 8 | 2
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.181, Regression, Logistic; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.03 to 13.55]
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.073, Regression, Logistic; Odds Ratio (OR) = 3.3, 95% CI 2-sided [0.90 to 12.13]
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.037, Regression, Logistic; Odds Ratio (OR) = 3.5, 95% CI 2-sided [1.08 to 11.48]
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.814, Regression, Logistic; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.40 to 3.25]

2. Primary Outcome: The Number of Participants With Adverse Events and Serious Adverse Events Following Administration of VIS410
Description: Safety and tolerability of 2 dose levels of a single intravenous (IV) dose of VIS410 when administered in combination with oseltamivir in hospitalized participants with influenza A infection. Data presents the count of participants who experienced an adverse event (AE) or serious treatment emergent adverse events (TEAE).
Time Frame: 56 days
Population: Safety Population: Included all ITT participants (participants who randomized to treatment) who received IV study drug. Participants were grouped according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 28 | 57 | 30
Participants
  Participants with adverse events | 16 | 22 | 38 | 16
  Participants with at least one serious treatment emergent adverse events | 6 | 4 | 10 | 6

3. Secondary Outcome: Time to Cessation of Oxygen Support Compared to Oseltamivir Alone Among Patients Requiring Supplemental Oxygen Therapy With Baseline Room Air <= 92%
Description: Time to cessation of O2 support in patients with supplemental oxygen with baseline room air <= 92%. Patients with treatment resulting in a stable SpO2 by pulse oximetry. Stable SpO2 is defined as two consecutive SpO2 values of >92% on room air that are at least 8 hours apart.
Time Frame: Baseline to Day 56
Population: Modified intent to treat population (MITT), number of participants who had cessation of oxygen support.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 18 | 15 | 33 | 15
Hours | 92.5 [45.5 to 138.7] | 101.3 [26.9 to 114.6] | 97.3 [45.5 to 124.7] | 79.0 [41.7 to 103.2]
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; The VIS410 high-dose group was compared against the placebo group. The null hypothesis was defined as no treatment difference; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.748, Chi-squared — p-value is not adjusted for multiple comparisons, which were performed at the 0.05 significance level. The goal will be used to assess the strength of evidence to select the endpoints for a Phase 3 trial; All statistical comparisons were performed using 2-sided tests at the 0.05 significance level
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; The VIS410 low-dose group was compared against the placebo group. The null hypothesis was defined as no treatment difference; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.940, Chi-squared — p-value is not adjusted for multiple comparisons, which were performed at the 0.05 significance level; All statistical comparisons were performed using 2-sided tests at the 0.05 significance level
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; The total VIS410 high-dose group (high-dose + low-dose) was compared against the placebo group. The null hypothesis was defined as no treatment difference; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.902, Chi-squared — p-value is not adjusted for multiple comparisons, which were performed at the 0.05 significance level; All statistical comparisons were performed using 2-sided tests at the 0.05 significance level
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; The VIS410 high-dose group was compared against the VIS410 low-dose group. The null hypothesis was defined as no treatment difference; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.283, Chi-squared — p-value is not adjusted for multiple comparisons, which were performed at the 0.05 significance level; All statistical comparisons were performed using 2-sided tests at the 0.05 significance level

4. Secondary Outcome: Time to Cessation of Oxygen Support for Any Patient Requiring Supplemental Oxygen Therapy
Description: Time to cessation of oxygen support in all patients with supplemental oxygen (regardless of oxygen saturation).
Time Frame: Baseline to Day 56
Population: Modified intent to treat population (MITT), number of participants who had cessation of oxygen support. NE = not estimable.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 27 | 26 | 53 | 25
Hours | 119.2 [82.3 to 257.0] | 129.7 [99.3 to NA] — Data are not estimable due to the insufficient number of participants with events for two main reasons. First measured baseline room air oxygen saturation was >92% in some subjects and in others the subject was already on supplemental oxygen and a measurement on room air at baseline was not obtained. | 124.7 [83.6 to NA] — Data are not estimable due to the insufficient number of participants with events for two main reasons. First measured baseline room air oxygen saturation was >92% in some subjects and in others the subject was already on supplemental oxygen and a measurement on room air at baseline was not obtained. | 112.2 [74.2 to NA] — Data are not estimable due to the insufficient number of participants with events for two main reasons. First measured baseline room air oxygen saturation was >92% in some subjects and in others the subject was already on supplemental oxygen and a measurement on room air at baseline was not obtained.
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.919, Chi-squared — p-value is not adjusted for multiple comparisons, which were performed at the 0.05 significance level; All statistical comparisons were performed using 2-sided tests at the 0.05 significance level
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.900, Chi-squared — p-value is not adjusted for multiple comparisons, which were performed at the 0.05 significance level; All statistical comparisons were performed using 2-sided tests at the 0.05 significance level
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; The combined VIS410 high- and low-dose groups was compared against the placebo group. The null hypothesis was defined as no treatment difference; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.990, Chi-squared — p-value is not adjusted for multiple comparisons; All statistical comparisons were performed using 2-sided tests at the 0.05 significance level
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; [analysis description as in outcome 3, analysis 4]; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.521, Chi-squared — The p-value is not adjusted for multiple comparisons; All statistical comparisons were performed using 2-sided tests at the 0.05 significance level

5. Secondary Outcome: Viral Titer in Upper Respiratory Samples by qRT-PCR
Description: The difference between VIS410 + oseltamivir and oseltamivir alone treatment groups in peak viral load by qRT-PCR from nasopharyngeal swabs through Day 14
Time Frame: Day 14
Population: The modified ITT (MITT) population included all participants who received IV study drug and were confirmed influenza A positive by qRT-PCR in central lab analysis of pre-dose Day 1 and/or post-dose Day 1. Participants were grouped according to the randomly assigned treatment. All efficacy analyses including the primary efficacy analyses were performed in the MITT population
Measure: Mean (Standard Deviation); unit: log10 virus particles/mL
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 27 | 27 | 54 | 28
log10 virus particles/mL | 6.479 (1.3860) | 6.378 (1.1320) | 6.429 (1.2544) | 6.169 (1.2489)
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.360, ANOVA — All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons

6. Secondary Outcome: Viral Nasopharyngeal AUC
Description: The difference between VIS410 + oseltamivir and oseltamivir alone treatment groups in nasopharyngeal qRT-PCR area under the viral load-time curve (AUC) from baseline to Day 5.
Time Frame: Day 1 Predose, Day 1 End of Infusion, Day 3, Day 5
Population: The modified ITT (MITT) population included all participants who received IV study drug and were confirmed influenza A positive by qRT-PCR in central lab analysis of pre-dose Day 1 and/or post-dose Day 1. Participants were grouped according to the randomly assigned treatment.
Measure: Mean (Standard Deviation); unit: Day*Log10 virus particles/ mL
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 27 | 27 | 54 | 28
Day*Log10 virus particles/ mL | 18.329 (6.7272) | 15.999 (4.9232) | 17.164 (5.9559) | 17.727 (5.9824)
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.735, ANOVA
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.259, ANOVA
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.644, ANOVA — The p-value is not adjusted for multiple comparisons. All statistical comparisons were performed using 2-sided tests at the 0.05 significance level
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.146, ANOVA

7. Secondary Outcome: Area Under the Viral Load-Time Curve (VL AUC) Based on qRT-PCR From Nasopharyngeal Swabs Through Day 7
Description: The difference between VIS410 + oseltamivir and oseltamivir alone treatment groups in nasopharyngeal qRT-PCR area under the viral load-time curve (AUC) from baseline to Day 7.
Time Frame: Day 1 Predose, Day 1 End of Infusion, Day 3, Day 5, Day 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Day*vp/mL
Groups:
- Total VIS410: Combined results from VIS410 high and low dose groups
Arm/Group | VIS410 High Dose | VIS410 Low Dose | Total VIS410 | Placebo
Number analyzed (Participants) | 27 | 27 | 54 | 27
Day*vp/mL | 25.490 (9.0440) | 22.394 (7.9006) | 23.942 (8.5550) | 24.337 (8.8837)
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.624, ANOVA — [p-value comment as in outcome 6, analysis 3]
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.399, ANOVA — [p-value comment as in outcome 6, analysis 3]
Statistical Analysis 3: Comparison: Total VIS410 vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.837, ANOVA
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.183, ANOVA

8. Secondary Outcome: Area Under the Viral Load-Time Curve (VL AUC) Based on qRT-PCR From Nasopharyngeal Swabs Through Day 14
Description: The difference between VIS410 + oseltamivir and oseltamivir alone treatment groups in nasopharyngeal qRT-PCR area under the viral load-time curve (AUC) from baseline to Day 14.
Time Frame: Day 1 Predose, Day 1 End of Infusion, Day 3, Day 5, Day 7, Day 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Day*vp/mL
Arm/Group | VIS410 High Dose | VIS410 Low Dose | Total VIS410 | Placebo
Number analyzed (Participants) | 26 | 26 | 52 | 25
Day*vp/mL | 37.356 (17.6513) | 35.172 (18.6217) | 36.264 (17.9980) | 36.668 (17.2015)
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.880, ANOVA
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.778, ANOVA
Statistical Analysis 3: Comparison: Total VIS410 vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.940, ANOVA
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.662, ANOVA

9. Secondary Outcome: Median Time to Resolution of Viral Load by Treatment Arm by qRT-PCR - From End of Infusion
Description: Number of days from the end of infusion until virus is no longer detectable (at or below the limit of detection) with no samples following that are greater than the BLQ through the Day 14 (quantitative reverse-transcription polymerase chain reaction - qRT-PCR)
Time Frame: 14 days
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | VIS410 High Dose | VIS410 Low Dose | Total VIS410 | Placebo
Number analyzed (Participants) | 27 | 27 | 54 | 28
Days | 13.5 [8.0 to 14.7] | 12.7 [5.9 to 13.7] | 12.7 [10.7 to 13.7] | 11.9 [6.5 to 13.7]
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; Test type: Other; p = 0.640, Chi-squared; A Wald Chi-square statistic from a Cox proportional model was used for comparisons of treatment groups
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; Test type: Other; p = 0.775, Chi-squared; A Wald Chi-square statistic from a Cox proportional model was used for comparisons of treatment groups
Statistical Analysis 3: Comparison: Total VIS410 vs Placebo; Test type: Other; p = 0.701, Chi-squared; A Wald Chi-square statistic from a Cox proportional model was used for comparisons of treatment groups
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; Test type: Other; p = 0.638, Chi-squared; A Wald Chi-square statistic from a Cox proportional model was used for comparisons of treatment groups

10. Secondary Outcome: Number of Participants in Whom Peak Viral Load Occurred Post Baseline Measured by qRT-PCR
Description: Number of participants in whom peak viral load is observed post-baseline based on quantitative reverse-transcription polymerase chain reaction (qRT-PCR). Post-baseline was considered the day 3 sample or later.
Time Frame: 14 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 28 | 57 | 28
Participants | 5 | 1 | 6 | 1
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; Test type: Other; p = 0.127, Regression, Logistic
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; Test type: Other; p = 1.000, Regression, Logistic
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; Test type: Other; p = 0.458, Regression, Logistic
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; Test type: Other; p = 0.127, Regression, Logistic

11. Secondary Outcome: Peak Viral Load by TCID50
Description: Peak viral load based on TCID50 from nasopharyngeal swabs
Time Frame: Day 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: log10 TCID50/mL
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 27 | 27 | 54 | 28
log10 TCID50/mL | 3.047 (2.1651) | 2.714 (1.7415) | 2.881 (1.9534) | 2.604 (2.0278)
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.371, ANOVA
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.735, ANOVA
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.476, ANOVA
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.581, ANOVA

12. Secondary Outcome: Number of Participants in Whom Peak Viral Load Occurred Post Baseline Measured by TCID50
Description: Number of participants in whom peak viral load occurred post-baseline measured by TCID50. Post-baseline was considered the day 3 sample or later.
Time Frame: 56 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 28 | 57 | 28
Participants | 1 | 0 | 1 | 1
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; Test type: Other; p = 0.980, Regression, Logistic
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; Test type: Other; p = 0.955, Regression, Logistic
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; Test type: Other; p = 0.955, Regression, Logistic
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; Test type: Other; p = 0.955, Regression, Logistic

13. Secondary Outcome: Viral Nasopharyngeal AUC by TCID50
Description: The area under the viral load-time curve (AUC) for VIS410 + oseltamivir and oseltamivir alone treatment groups from baseline to Day 5 measured by TCID50 from nasopharyngeal swabs.
Time Frame: 5 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Day*TCID50 log10/ml
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 27 | 27 | 54 | 28
Day*TCID50 log10/ml | 3.826 (4.2581) | 2.823 (2.4121) | 3.324 (3.4649) | 3.519 (3.5317)
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.695, ANOVA
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.542, ANOVA
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.899, ANOVA
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.321, ANOVA

14. Secondary Outcome: Viral Nasopharyngeal AUC by TCID50
Description: The area under the viral load-time curve (AUC) for VIS410 + oseltamivir and oseltamivir alone treatment groups from baseline to Day 7 measured by TCID50 from nasopharyngeal swabs.
Time Frame: 7 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Day*TCID50 log10/ml
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 27 | 27 | 54 | 27
Day*TCID50 log10/ml | 4.140 (5.2238) | 2.886 (2.5260) | 3.513 (4.1131) | 3.711 (4.2207)
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.663, ANOVA
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.540, ANOVA
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.918, ANOVA
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.294, ANOVA

15. Secondary Outcome: Negative Viral Cultures by Study Day
Description: Number of participants negative for viral titer by study day determined by TCID50 on nominal days 3, 5, 7
Time Frame: Nominal days 3, 5, 7
Population: The modified ITT (MITT) population included all participants who received IV study drug and were confirmed influenza A positive by qRT-PCR in central lab analysis of pre-dose Day 1 and/or post-dose Day 1. Participants were grouped according to the randomly assigned treatment, who also had a positive baseline viral culture based on TCID50.
Measure: Count of Participants; unit: Participants
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 28 | 57 | 28
Participants
  Participants with negative viral cultures by Day 3. | 23 | 24 | 47 | 19
  Participants with negative viral cultures by Day 5.: number analyzed (Participants) | 27 | 27 | 54 | 28
  Participants with negative viral cultures by Day 5. | 25 | 26 | 51 | 25
  Participants with negative viral cultures by Day 7.: number analyzed (Participants) | 28 | 27 | 55 | 27
  Participants with negative viral cultures by Day 7. | 28 | 27 | 55 | 27

16. Secondary Outcome: Median Time to Resolution of Viral Load by Treatment Arm by TCID50 - From End of Infusion
Description: Number of days from the end of infusion until virus is no longer detectable (at or below the limit of detection) with no samples following that are greater than the BLQ through the Day 7 (TCID50)
Time Frame: 7 Days
Population: The modified ITT (MITT) population included all participants who received IV study drug and were confirmed influenza A positive by TCID50 in central lab analysis of pre-dose Day 1 and/or post-dose Day 1. Participants were grouped according to the randomly assigned treatment, who also had a positive baseline viral culture based on TCID50.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 27 | 27 | 54 | 27
Days | 1.7 [0.6 to 1.9] | 1.7 [1.5 to 1.8] | 1.7 [1.6 to 1.7] | 1.8 [0.0 to 2.5]
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.250, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.133, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.177, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.360, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups

17. Secondary Outcome: Median Time to Resolution of Viral Load by Treatment Arm by TCID50 - From Onset of Symptoms
Description: Number of days from the onset of symptoms until virus is no longer detectable (at or below the limit of detection) with no samples following that are greater than the BLQ through the Day 7 (TCID50)
Time Frame: 7 Days
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 27 | 27 | 54 | 27
Days | 4.7 [3.6 to 5.3] | 4.8 [3.9 to 5.1] | 4.8 [4.1 to 4.9] | 4.4 [4.0 to 5.7]
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.636, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.446, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.530, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.463, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups

18. Secondary Outcome: Time to Clinical Response (4 Out of 5 Vital Signs)
Description: Median time to clinical response defined by resolution of at least 4 of 5 vital signs:
  * Afebrile with core temperature ≤ 37.8°C, without use of antipyretics (oral ≤ 37.2°C)
  * Oxygen saturation ≥ 95% on room air without support or a return to preinfection status, if pre-infection status was < 95%
  * Pulse rate ≤ 100/min
  * Systolic blood pressure ≥ 90 mm/Hg, without vasopressor use
  * Respiratory rate ≤ 24 beats per minute
Time Frame: Day 56
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 27 | 56 | 26
hours | 2.6 [2.2 to 21.9] | 2.6 [2.2 to 24.0] | 2.6 [2.2 to 21.9] | 2.8 [2.2 to 44.2]
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.152, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.176, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.157, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.844, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups

19. Secondary Outcome: Time to Complete Clinical Response (Resolution of All Vital Signs)
Description: Median time to clinical response defined by resolution of at all 5 vital signs:
  * Afebrile with core temperature ≤ 37.8°C, without use of antipyretics (oral ≤ 37.2°C)
  * Oxygen saturation ≥ 95% on room air without support or a return to pre-infection status, if pre-infection status was < 95%
  * Pulse rate ≤ 100/min
  * Systolic blood pressure ≥ 90 mm/Hg, without vasopressor use
  * Respiratory rate ≤ 24 beats per minute
Time Frame: Day 56
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 25 | 24 | 49 | 22
hours | 103.0 [45.4 to 170.6] | 114.6 [47.5 to 166.1] | 103.0 [47.5 to 170.6] | 99.8 [63.0 to 168.5]
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.531, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.582, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.550, Chi-squared; Wald Chi-square statistic from a Cox proportional model is used for comparisons of treatment groups
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.840, Chi-squared; P-value determined based on Cox proportional hazards model Wald Chi-Square Statistic

20. Secondary Outcome: Clinical Status Ordinal Scale Mean Area Under the Curve Through Day 7
Description: Summary of area under the curve (AUC) over time for seven-level ordinal scale. Area under the curve (AUC) is calculated using the linear trapezoidal rule. Seven-Level Ordinal Scale is a hierarchical scale with the classifications presented from the worst clinical outcome to the best clinical outcome in descending order with 7=death, 6=Intensive care unit (ICU) stay with mechanical ventilation , 5=ICU stay without mechanical ventilation, 4=Non-ICU hospitalization with supplemental oxygen, 3=Non-ICU hospitalization without supplemental oxygen, 2=Discharge with partial resumption of normal activities, 1=Discharge with full resumption of normal activities. Time frame is from baseline to day 7. Therefore, maximum and minimum values possible for the AUC Clinical Status Ordinal Scale scores range from 7 to 49.
Time Frame: Baseline to Day 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: day*units on a scale
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 28 | 57 | 28
day*units on a scale | 23.6 (5.55) | 22.4 (7.47) | 23.0 (6.53) | 21.4 (4.97)
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.3534, ANCOVA
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.7839, ANCOVA
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.4893, ANCOVA
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.5101, ANCOVA

21. Secondary Outcome: Clinical Status Ordinal Scale Mean Area Under the Curve Through Day 14.
Description: Summary of area under the curve (AUC) over time for seven-level ordinal scale. Area under the curve (AUC) is calculated using the linear trapezoidal rule. Seven-Level Ordinal Scale is a hierarchical scale with the classifications presented from the worst clinical outcome to the best clinical outcome in descending order with 7=death, 6=Intensive care unit (ICU) stay with mechanical ventilation , 5=ICU stay without mechanical ventilation, 4=Non-ICU hospitalization with supplemental oxygen, 3=Non-ICU hospitalization without supplemental oxygen, 2=Discharge with partial resumption of normal activities, 1=Discharge with full resumption of normal activities. Time frame is from baseline to day 14. Therefore, maximum and minimum values possible for the AUC Clinical Status Ordinal Scale scores range from 14 to 98.
Time Frame: Baseline to Days 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: day*units on a scale
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 28 | 57 | 28
day*units on a scale | 40.3 (15.21) | 38.2 (18.73) | 39.3 (16.91) | 35.8 (12.54)
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.5436, ANCOVA
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.8215, ANCOVA
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.6319, ANCOVA
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.7011, ANCOVA

22. Secondary Outcome: Comparison of Clinical Status on Seven-level Ordinal Scale Scores
Description: Summary of Clinical Outcome on Seven-Level Ordinal Scale through Day 14. Worst post-baseline assessment observed.
  Seven-Level Ordinal Scale is a hierarchical scale with the classifications presented from the worst clinical outcome to the best clinical outcome in descending order with 7=death, 6=Intensive care unit (ICU) stay with mechanical ventilation , 5=ICU stay without mechanical ventilation, 4=Non-ICU hospitalization with supplemental oxygen, 3=Non-ICU hospitalization without supplemental oxygen, 2=Discharge with partial resumption of normal activities, 1=Discharge with full resumption of normal activities.
Time Frame: Day 14
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 28 | 57 | 28
Participants
  Death | 1 | 2 | 3 | 1
  ICU stay with mechanical ventilation | 4 | 2 | 6 | 2
  ICU stay without mechanical ventilation | 4 | 5 | 9 | 3
  Non-ICU hospitalization with supplemental oxygen | 18 | 17 | 35 | 20
  Non-ICU hospitalization without supplemental oxygen | 2 | 1 | 3 | 2
  Discharge with partial resumption of normal activities | 0 | 1 | 1 | 0
  Discharge with full resumption of normal activities | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: VIS410 High Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.478, Regression, Logistic
Statistical Analysis 2: Comparison: VIS410 Low Dose vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.468, Regression, Logistic
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.412, Regression, Logistic
Statistical Analysis 4: Comparison: VIS410 High Dose vs VIS410 Low Dose; All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Test type: Superiority — The null hypothesis was defined as no treatment difference; p = 0.982, Regression, Logistic

23. Secondary Outcome: Total Number of Days on Ventilation
Description: Total number of days on ventilation for participants who used ventilation, including participants on ventilation at baseline
Time Frame: 56 days
Population: Participants requiring ventilation from the mITT population. The modified ITT (MITT) population included all participants who received IV study drug and were confirmed influenza A positive by qRT-PCR in central lab analysis of pre-dose Day 1 and/or post-dose Day 1. Participants were grouped according to the randomly assigned treatment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 5 | 3 | 8 | 3
days | 5.2 (4.55) | 7.0 (5.20) | 5.9 (4.52) | 11.7 (7.51)

24. Secondary Outcome: Comparison of Ordinal Scale Parameters - Days on Ventilation
Description: Total number of days on ventilation for participations who used ventilation, including participants on ventilation at baseline. Better and worse outcome groups defined based on the Seven-Level Ordinal Scale scores, "<= 4 Seven-Level Ordinal Scale Score" is better; "> 4 Seven-Level Ordinal Scale Score" is worse group.
  Seven-Level Ordinal Scale is a hierarchical scale with the classifications presented from the worst clinical outcome to the best clinical outcome in descending order with 7=death, 6=Intensive care unit (ICU) stay with mechanical ventilation , 5=ICU stay without mechanical ventilation, 4=Non-ICU hospitalization with supplemental oxygen, 3=Non-ICU hospitalization without supplemental oxygen, 2=Discharge with partial resumption of normal activities, 1=Discharge with full resumption of normal activities.
Time Frame: 56 days
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: days
Arm/Group | VIS410 High Dose | VIS410 Low Dose | Total VIS410 | Placebo
Number analyzed (Participants) | 5 | 3 | 8 | 3
days
  > 4 Seven-Level Ordinal Scale Score: number analyzed (Participants) | 5 | 3 | 8 | 2
  > 4 Seven-Level Ordinal Scale Score | 5.2 (4.55) | 7.0 (5.2) | 5.9 (4.52) | 8.0 (5.66)
  <= 4 Seven-Level Ordinal Scale Score: number analyzed (Participants) | 0 | 0 | 0 | 1
  <= 4 Seven-Level Ordinal Scale Score |  |  |  | 19.0 (NA) — There is only 1 participant analyzed.

25. Secondary Outcome: Total Number of Days in ICU
Description: Total number of days in intensive care (ICU) for participants who admitted to the ICU, including participants in ICU at baseline
Time Frame: 56 days
Population: Participants admitted to the ICU from the mITT population. The modified ITT (MITT) population included all participants who received IV study drug and were confirmed influenza A positive by qRT-PCR in central lab analysis of pre-dose Day 1 and/or post-dose Day 1. Participants were grouped according to the randomly assigned treatment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 11 | 10 | 21 | 5
days | 8.5 (7.43) | 6.8 (3.71) | 7.7 (5.88) | 14.0 (9.38)

26. Secondary Outcome: Comparison of Ordinal Scale Parameters - Days in ICU
Description: Total number of days in intensive care for participants who admitted to ICU, including participants in ICU at baseline. Better and worse outcome groups defined based on the Seven-Level Ordinal Scale scores, "<= 4 Seven-Level Ordinal Scale Score" is better; "> 4 Seven-Level Ordinal Scale Score" is worse group.
  Seven-Level Ordinal Scale is a hierarchical scale with the classifications presented from the worst clinical outcome to the best clinical outcome in descending order with 7=death, 6=Intensive care unit (ICU) stay with mechanical ventilation , 5=ICU stay without mechanical ventilation, 4=Non-ICU hospitalization with supplemental oxygen, 3=Non-ICU hospitalization without supplemental oxygen, 2=Discharge with partial resumption of normal activities, 1=Discharge with full resumption of normal activities.
Time Frame: 56 days
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: days
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 11 | 10 | 21 | 5
days
  > 4 Seven-Level Ordinal Scale Score: number analyzed (Participants) | 11 | 10 | 21 | 4
  > 4 Seven-Level Ordinal Scale Score | 8.5 (7.43) | 6.8 (3.71) | 7.7 (5.88) | 10.8 (6.85)
  <= 4 Seven-Level Ordinal Scale Score" is better: number analyzed (Participants) | 0 | 0 | 0 | 1
  <= 4 Seven-Level Ordinal Scale Score" is better |  |  |  | 27.0 (NA) — There is only 1 participant analyzed.

27. Secondary Outcome: Number of Days to Resumption of Usual Activities
Description: Number of days until resumption of usual activities by treatment group
Time Frame: Day 56
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: days
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 28 | 57 | 28
days | 11.9 (3.07) | 10.3 (4.10) | 11.1 (3.67) | 11.5 (3.38)

28. Secondary Outcome: All Cause and Attributable Mortality at Day 14
Description: Number of patients experiencing all-cause and attributable mortality rates at Day 14. Attributable mortality was derived from the Complication of Influenza eCRF; all-cause mortality was derived from Complication of Influenza, Seven-Level Ordinal Scale, AE and Study Completion eCRFs
Time Frame: Day 14
Population: The safety population included all ITT participants who received IV study drug. Participants were grouped according to the actual treatment received.
Measure: Number; unit: participants
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 29 | 58 | 30
participants
  All-cause mortality Day 14 | 1 | 2 | 3 | 1
  Attributable mortality Day 14 | 1 | 2 | 3 | 1

29. Secondary Outcome: All Cause and Attributable Mortality by Day 28
Description: Number of patients experiencing all-cause and attributable mortality by Day 28. Attributable mortality was derived from the Complication of Influenza eCRF; all-cause mortality was derived from Complication of Influenza, Seven-Level Ordinal Scale, AE and Study Completion eCRFs
Time Frame: Day 28
Population: as for outcome 28
Measure: Number; unit: participants
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 29 | 58 | 30
participants
  All-cause mortality Day 28 | 1 | 2 | 3 | 2
  Attributable mortality Day 28 | 1 | 2 | 3 | 2

30. Secondary Outcome: All Cause and Attributable Mortality Day 56
Description: Number of patients experiencing all-cause and attributable mortality by Day 56. Attributable mortality was derived from the Complication of Influenza eCRF; all-cause mortality was derived from Complication of Influenza, Seven-Level Ordinal Scale, AE and Study Completion eCRFs
Time Frame: Day 56
Population: as for outcome 28
Measure: Number; unit: participants
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 29 | 58 | 30
participants
  All-cause mortality Day 56 | 1 | 2 | 3 | 2
  Attributable mortality Day 56 | 1 | 2 | 3 | 2

31. Secondary Outcome: Healthcare Resource Utilization. Days in Hospital and/or ICU
Description: Total number of days in hospital and/or ICU from admission to discharge
Time Frame: Day 56
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 28 | 57 | 28
Days | 11.4 (8.6) | 9.6 (7.02) | 10.5 (7.84) | 9.6 (6.38)

32. Secondary Outcome: Comparison of Ordinal Scale Parameters - Days in Hospital/ICU
Description: Total number of days in hospital or intensive care for participations who were admitted to Hospital/ICU, including participants in Hospital/ICU at baseline. Better and worse outcome groups defined based on the Seven-Level Ordinal Scale scores, "<= 4 Seven-Level Ordinal Scale Score" is better; "> 4 Seven-Level Ordinal Scale Score" is worse group.
  Seven-Level Ordinal Scale is a hierarchical scale with the classifications presented from the worst clinical outcome to the best clinical outcome in descending order with 7=death, 6=Intensive care unit (ICU) stay with mechanical ventilation , 5=ICU stay without mechanical ventilation, 4=Non-ICU hospitalization with supplemental oxygen, 3=Non-ICU hospitalization without supplemental oxygen, 2=Discharge with partial resumption of normal activities, 1=Discharge with full resumption of normal activities.
Time Frame: 56 days
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: days
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 28 | 57 | 28
days
  > 4 Seven-Level Ordinal Scale Score: number analyzed (Participants) | 11 | 10 | 21 | 4
  > 4 Seven-Level Ordinal Scale Score | 15.9 (12.47) | 12.6 (9.08) | 14.3 (10.85) | 13.8 (9.74)
  <= 4 Seven-Level Ordinal Scale Score: number analyzed (Participants) | 18 | 18 | 36 | 24
  <= 4 Seven-Level Ordinal Scale Score | 8.6 (3.01) | 7.9 (5.13) | 8.3 (4.16) | 8.9 (5.64)

33. Secondary Outcome: Number of Participants With Rehospitalization Due to Relapse
Description: Number of participants with rehospitalization due to influenza A relapse
Time Frame: Day 56
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 28 | 57 | 28
Participants
  Rehospitalization due to relapse--Yes | 2 | 1 | 3 | 3
  Rehospitalization due to relapse--No | 27 | 27 | 54 | 25

34. Secondary Outcome: Number of Participants With Influenza-related Complications
Description: Summary of influenza symptom complications, including baseline and incident complications
Time Frame: Day 56
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 29 | 28 | 57 | 28
Participants
  Participants with at least 1 complication of Influenza | 4 | 4 | 8 | 4
  Participants with pneumonia | 3 | 1 | 4 | 0
  Participants with sinusitis | 0 | 1 | 1 | 0
  Other chronic pulmonary disease | 0 | 0 | 0 | 2
  Death | 1 | 2 | 3 | 2
  Bacterial pneumonia | 3 | 1 | 4 | 0

35. Secondary Outcome: The Maximum Concentration (Cmax) of VIS410 in Participant's Serum
Description: Summary of Serum VIS410 Pharmacokinetic Parameters in PK Population by maximum concentration (Cmax) of VIS410 in participant's serum.
Time Frame: Baseline, end of infusion, Day 5, Day 14, Day 28, Day 56
Population: The PK population included all participants who received IV study drug and had at least 1 PK parameter that could be calculated.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | VIS410 High Dose | VIS410 Low Dose
Number analyzed (Participants) | 27 | 28
µg/mL | 1301.037 (241.0838) | 786.393 (202.7963)

36. Secondary Outcome: The Area Under the Concentration/Time Curve of VIS410 in Participant's Serum
Description: Summary of Serum VIS410 Pharmacokinetic Parameters in PK Population by the area under the concentration/time curve from 0 to infinity (AUC0-inf) of VIS410 in participant's serum.
Time Frame: Baseline, end of infusion, Day 5, Day 14, Day 28, Day 56
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | VIS410 High Dose | VIS410 Low Dose
Number analyzed (Participants) | 23 | 27
day*µg/mL | 11326.522 (4205.1144) | 6934.815 (2304.3093)

37. Secondary Outcome: The Clearance Rate (Cl) of VIS410 in Participant's Serum
Description: Summary of Serum VIS410 Pharmacokinetic Parameters in PK Population by the clearance rate (Cl) of VIS410 in participant's serum.
Time Frame: PK samples were collected on days 1, 5, 14, 28 and 56.
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | VIS410 High Dose | VIS410 Low Dose
Number analyzed (Participants) | 23 | 27
mL/day | 401.652 (143.6763) | 325.926 (137.6743)

38. Secondary Outcome: The Half-life of VIS410 in Participant's Serum
Description: Summary of Serum VIS410 Pharmacokinetic Parameters in PK Population by the half-life (t1/2) of VIS410 in participant's serum.
Time Frame: PK samples were collected on days 1, 5, 14, 28 and 56.
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | VIS410 High Dose | VIS410 Low Dose
Number analyzed (Participants) | 23 | 27
mL/day | 9.407 (3.5549) | 9.839 (3.2465)

39. Secondary Outcome: Anti-VIS410 Antibody Testing
Description: Summary of the maximum fold increase for anti-VIS410 antibody testing for VIS410 groups and placebo.
Time Frame: From anti-VIS410 antibody samples collected on days 28 and 56.
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 25 | 26 | 51 | 25
Participants
  1 to 4 fold | 22 | 24 | 46 | 25
  >4 to 16 fold | 2 | 1 | 3 | 0
  >16 to 64 fold | 1 | 0 | 1 | 0
  >64 fold | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events for 55 days following dosing of VIS410 or placebo.
Description: Each adverse event was graded on a 4-point scale (Grades 1-4) of increasing intensity according to the Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table.
Arm/Group | VIS410 High Dose | VIS410 Low Dose | Total VIS410 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/29 | 2/29 | 3/58 | 3/30
Serious Adverse Events (participants affected / at risk) | 7/29 | 6/29 | 13/58 | 9/30
Other Adverse Events (participants affected / at risk) | 11/29 | 13/29 | 24/58 | 7/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VIS410 High Dose (N=29) | VIS410 Low Dose (N=29) | Total VIS410 (N=58) | Placebo (N=30)
Cardiac Arrest (Cardiac disorders) | 1 | 2 | 3 | 3
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 1 | 0
Septic encephalopathy (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VIS410 High Dose (N=29) | VIS410 Low Dose (N=29) | Total VIS410 (N=58) | Placebo (N=30)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 9 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 6 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Pneumonia (Infections and infestations) | 3 | 1 | 4 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4 | 2
Hypertension (Vascular disorders) | 2 | 2 | 4 | 3

LIMITATIONS AND CAVEATS:
Approximately 120 participants were planned to be included in the study. A total of 89 participants were randomized to treatment of which 73 subjects completed the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution may not publish study results until publication of the results of the full study or 2 years after study completion.

The institution must provide a copy of any proposed publication to the Sponsor at least 40 days in advance

The Sponsor may:

1. provide comments on the proposed publication;
2. request delay of the publication for 120 days;
3. request that specified confidential information be removed

DOCUMENTS (2):
  • Study Protocol (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT03040141/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT03040141/SAP_001.pdf